CLINICAL TRIAL: NCT04712409
Title: Characterization of Intestinal Hormone and Glucose Dynamics to Unravel the Antidiabetic Effect of Bariatric Surgery
Brief Title: Surgical Innovation for Diabetes Treatment 2
Acronym: SURIDIAB2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Sao Sebastiao (Other)
Collaborators: Instituto de Ciências Biomédicas Abel Salazar (Other); The Novo Nordisk Foundation Center for Basic Metabolic Research (Other)
Responsible Party: Principal Investigator, Marta Guimarães, Principal Investigator, Hospital de Sao Sebastiao
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSS
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Enteroendocrine Physiological Changes in Superobese Patients Submitted to Two Different Bariatric Procedures; Determine Whether BPD With DS or SADI-S as Primary or Revisional Surgery is Superior Than the Other as First Choice for the Superobese; Determine Whether or Not Revision Surgery is as Effective as Primary Surgery and Understand the Physiological Mechanisms Inherent in These Putative Differences
Keywords: Bariatric Surgery; Superobesity; Revisional Bariatric Surgery; Single anastomosis duodeno-ileal bypass; Biliopancreatic diversion with duodenal switch
MeSH Terms: interventions — Biliopancreatic Diversion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SADI-S as a primary surgery (Active Comparator)
  Interventions: Procedure: Single anastomosis duodeno-ileal bypass
- BPD-DS as a primary surgery (Active Comparator)
  Interventions: Procedure: Biliopancreatic diversion with duodenal switch
- SADI-S as a revisional procedure (Active Comparator)
  Interventions: Procedure: SADI-S as a revisional procedure
- BPD-DS as a revisional procedure (Active Comparator)
  Interventions: Procedure: BPD-DS as a revisional procedure

INTERVENTIONS:
Procedure: Single anastomosis duodeno-ileal bypass — Sleeve gastrectomy followed by division of the duodenum bypassing the jejunum with end-to-side duodeno-ileal diversion
  Other Names: SADI-S
  Arms: SADI-S as a primary surgery
Procedure: Biliopancreatic diversion with duodenal switch — Sleeve gastrectomy, followed by division of the duodenum bypassing the jejunum with end-to-side duedeno-ileal diversion and Roux-en-y entero-enteric anastomosis, leaving 100 cm common channel.
  Other Names: BPD-DS
  Arms: BPD-DS as a primary surgery
Procedure: SADI-S as a revisional procedure — In patients previously submitted to sleeve gastrectomy a single anastomosis duodeno-ileal bypass will be performed as 2nd time surgery
  Arms: SADI-S as a revisional procedure
Procedure: BPD-DS as a revisional procedure — In patients previously submitted to sleeve gastrectomy a biliopancreatic diversion with duodenal switch will be performed as 2nd time surgery
  Arms: BPD-DS as a revisional procedure

SUMMARY:
This study aims to understand the enteroendocrine physiological changes in superobese patients submitted to two different bariatric procedures (biliopancreatic diversion with duodenal switch versus single anastomosis duodeno-ileal bypass), when perfomed as primary or revisional surgeries (after a sleeve gastrectomy). The main purpose is to establish the metabolic changes obtained with the sleeve gastrectomy and how the revisional procedure maximizes those changes. Additionally, the study will determine whether BPD with DS or SADI-S is superior than the other as first choice for the superobese.

The study will monitor the enteroendocrine function before and after the ingestion of a mixed meal, in pre-operatory and post-surgery timepoints, comparing both primary and revisional surgeries.

DETAILED DESCRIPTION:
Abstract Obesity is a chronic disease whose global incidence keeps rising as the twenty first century goes on. Nowadays, the surgical approach constitutes the best treatment option for these patients, making the sleeve gastrectomy and the gastric bypass the more frequently performed bariatric surgeries.

However, the superobese patients (IMC≥ 50kg/m2) present variable weight loss resistance to the previous techniques, showing better results when submitted to disabsorptive procedures, namely the biliopancreatic diversion with duodenal switch, and the more recently created single anastomosis duodeno-ileal bypass. Each constitutes a revisional surgery option after a primary sleeve gastrectomy, reducing surgical and anesthesia risks. This has brought to light that some superobese patients do not need the revisional procedure as they achieve the weight loss target solely by the vertical gastrectomy.

Supported on the investigators' previous work and extensive experience performing both techniques, they now aim to understand the enteroendocrine physiological changes which each procedure accomplishes and compare them in terms of therapeutic efficacy among the superobese. The utmost goals will be to unravel the advantages of BPD-DS and SADI-S as primary or revisional surgeries, the differences between patients that respond well to sleeve gastrectomy alone and those who do not, and, finally, providing further insights on which procedure should be favoured over the other based on the patient characteristics.

Study Overview:

Participants in this study will have been submitted to either BPD-DS or SADI-S, as a primary or as a revisional surgery.

* Participants visits will be scheduled before surgery and after surgery at 3, 6 , 12 and 24 months for those who receive BPD-DS or SADI-S as a primary procedure.
* Those who are firstly submitted to the sleeve gastrectomy, visits will be scheduled before surgery and after surgery at 3 , 6 and 12 months. The revisional surgery will take place 1 year after the sleeve, with visits scheduled before surgery and after surgery at 3, 6 and 12 months.

In all these visits, detailed participants assessment will include vitals, anthropometric and biochemical evaluation, and the performance of a MMTT with plasma sampling for hormonal profiles. Intraoperative sampling of visceral and subcutaneous adipose tissue will take place during BPD-DS or SADI-S as a primary procedure and during the sleeve gastrectomy and repeated 1 year after the revisional surgery, either BPD-DS or SADI-S, is performed.

Participant Enrolment:

Participants will be selected from the cohort of patients referred for multidisciplinary evaluation by the clinical team for surgical treatment of obesity of the Centro Hospitalar Entre Douro e Vouga (CHEDV). Participants found to be suitable according to the entry criteria and who have accepted to participate will be enrolled in the study and assigned to one of the four study groups according to participants clinical features.

ELIGIBILITY:
Inclusion Criteria:

Bariatric surgery candidates

* BMI between 45 and 55 kg/m2
* Aged between 18 and 65 years at surgery

Exclusion Criteria:

* Previous abdominal surgery
* Diabetic patients (Hb A1c > 5,7%) prior to the bariatric procedure
* Treatment with antidiabetic drugs, except for purposes other than diabetes treatment, prior to the bariatric procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-16 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in body mass index | From enrolment to 12 months post-intervention in 4 visits: preoperative, 3, 6 and 12 months post-surgery
  Body mass index (BMI) combines height (in meters) and weight (in kilograms) and is calculated as weight over (height)^2. Therefore, it will be reported in kg/m^2. This parameter will be determined at each study timepoint (pre-operatory, 3, 6 and 12 months post-surgery) at presential visits to the clinic.
Change in glycated haemoglobin | From enrolment to 12 months post-intervention in 4 visits: preoperative, 3, 6 and 12 months
  Glycated haemoglobin (HbA1c) will be measured in percentage (%). This parameter will be assessed at each study timepoint (pre-operatory, 3, 6 and 12 months post- surgery) through routine complete biochemical evaluation.
Change in glucose dynamic profile | From enrolment to 12 months post-intervention in 4 visits: preoperative, 3, 6 and 12 months
  Glucose will be measured in mmol/L. This parameter will be assessed at each study timepoint (pre-operatory, 3, 6 and 12 months post-surgery) under fasting conditions and during a mixed-meal tolerance teste (MMTT) with blood collection at eight timed intervals (-10, 0, 15, 30, 45, 60, 90 and 120 minutes).
Change in insulin dynamic profile | From enrolment to 12 months post-intervention in 4 visits: preoperative, 3, 6 and 12 months post-surgery
  Insulin will be measured in mIU/L. This parameter will be assessed at each study timepoint (pre-operatory, 3, 6 and 12 months post-surgery) under fasting conditions and during a mixed-meal tolerance teste (MMTT) with blood collection at eight timed intervals (-10, 0, 15, 30, 45, 60, 90 and 120 minutes).
Change in glucagon dynamic profile | From enrolment to 12 months post-intervention in 4 visits: preoperative, 3, 6 and 12 months post-surgery
  Glucagon will be measured in pmol/L. This parameter will be assessed at each study timepoint (pre-operatory, 3, 6 and 12 months post-surgery) under fasting conditions and during a mixed-meal tolerance teste (MMTT) with blood collection at eight timed intervals (-10, 0, 15, 30, 45, 60, 90 and 120 minutes).
Change in GLP-1 dynamic profile | From enrolment to 12 months post-intervention in 4 visits: preoperative, 3, 6 and 12 months post-surgery
  Glucagon-like peptide-1 (GLP-1) will be measured in pmol/L. This parameter will be assessed at each study timepoint (pre-operatory, 3, 6 and 12 months post-surgery) under fasting conditions and during a mixed-meal tolerance teste (MMTT) with blood collection at eight timed intervals (-10, 0, 15, 30, 45, 60, 90 and 120 minutes).
Change in GIP dynamic profile | From enrolment to 12 months post-intervention in 4 visits: preoperative, 3, 6 and 12 months post-surgery
  Glucose-dependent insulinotropic polypeptide (GIP) will be measured in pmol/L. This parameter will be assessed at each study timepoint

SECONDARY OUTCOMES:
Hypertension remission rates | From enrolment to 12 months post-intervention in 4 visits: preoperative, 3, 6 and 12 months post-surgery
Dyslipidemia remission rates | From enrolment to 12 months post-intervention in 4 visits: preoperative, 3, 6 and 12 months post-surgery
Sleep Apnea remission rates | From enrolment to 12 months post-intervention in 4 visits: preoperative, 3, 6 and 12 months post-surgery
Metabolic syndrome remission rates | From enrolment to 12 months post-intervention in 4 visits: preoperative, 3, 6 and 12 months post-surgery

OTHER OUTCOMES:
Surgical morbidity | From surgery date to 3 months post-surgery
Surgical mortality | From surgery date to 3 months post-surgery
Late morbidity | From 3 months until 4 years post-surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Portugal (2):
  - São Sebastião Hospital, Santa Maria da Feira, Aveiro District
  - Hospital de São Sebastião, Santa Maria da Feira

IPD SHARING:
Plan to Share IPD: No